CLINICAL TRIAL: NCT03878290
Title: RiSE to Prevent Cardiovascular Disease in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Karen Saban, Associate Professor, Niehoff School of Nursing, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 210130
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Atherosclerosis; Stress; Hypertension; Dyslipidemias; Obesity; Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Hypertension; Dyslipidemias; Obesity; Diabetes Mellitus; Coronary Artery Disease | interventions — Ethnicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-week RiSE (Experimental): Participate in 8-week Resilience, Stress, and Ethnicity (RiSE) group based stress reduction program in which participants meet every week for approximately 2 hours for 8 consecutive weeks.
  Interventions: Behavioral: Resilience, Stress, and Ethnicity (RiSE)
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Resilience, Stress, and Ethnicity (RiSE) — Group based stress reduction program focused on helping minorities develop coping and empowerment skills
  Other Names: RiSE
  Arms: 8-week RiSE

SUMMARY:
The purpose of this pilot study is to evaluate an innovative 8-wk stress reduction program called Resilience, Stress and Ethnicity (RiSE) program designed to reduce chronic stress associated with perceived discrimination among African Americans. African Americans residing in the Maywood community between the ages of 25 and 75 with at least one cardiovascular disease risk factor such as being overweight, having high blood pressure, or diabetes will be enrolled. The following specific aims will be addressed:

Aim 1: Determine the feasibility and acceptability of the program as a strategy to reduce chronic stress in African Americans within the Maywood and surrounding community.

Aim 2: Examine the extent to which training in RiSE (1) improves psychological well being, (2) decreases inflammatory burden, and (3) reduces cardiovascular risk in African Americans

Participants will be randomized to either the RiSE program or the control (no intervention group). Participants will provide blood and saliva samples as well as complete written questionnaires asking them questions about their health, well-being, and early life at the start of the study, half way through the study (at 4 weeks), at the completion of the intervention (8 weeks) and 3 months after the completion of the intervention).

DETAILED DESCRIPTION:
The purpose of this study is to examine an 8-week stress reduction program for African Americans. The aim of this study is to determine the effectiveness of this stress reduction program in improving well-being and reducing risk for heart disease and stroke in African Americans.

No drugs are involved with this study. Participants will be randomized (randomly selected) to either participate in an 8 -week stress reduction program or a control group (no stress reduction program). The stress reduction program entails attending a 2- hour small group class once a week for 8 consecutive weeks at Loyola University in Maywood. Classes will be offered in the evening and will focus on teaching effective strategies for coping with daily stress, particularly stress associated with being an African American.

Blood and saliva samples will be collected at the beginning of the study, in the middle of the program (4 weeks), at the end of the program (8 weeks) and 3 months after the program ends. Blood samples will be analyzed for cholesterol levels, hemoglobin A1c (a measure that reflects blood sugar over time), and cytokines (which reflect inflammation in the body). Saliva samples will be assessed for a hormone called cortisol..

Participants will also complete several written questionnaires to gather information about their stress, social status, perceive discrimination, mood, diet and exercise. Participants will be paid $25 for each of the three data collection time points ($75 total). Those participants who are randomized to attend the stress reduction classes will also be provided $15 for each class that they attend (8 X $15 = $120) to help cover travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Living in Maywood community or surrounding area
* Able to speak, read, write English
* Have at least one of the following:
* Body Mass Index (BMI) > 25 (overweight or obese)
* Total cholesterol > 240
* Diabetes mellitus
* Systolic blood pressure the same or greater than 120 mmHg or diagnosis of hypertension and/or taking antihypertensive medication
* Atrial fibrillation
* Parental history of myocardial infarction (MI) (heart attack) prior to age 60

Exclusion Criteria:

* Current smoker (smoked in last month)
* History of myocardial infarction or ischemic heart disease
* Current cancer
* Active infection
* Major Immune-related disorder (lupus,MS)
* Substance abuse
* Immune-altering drugs
* Recent dental procedure (within past 72 hours
* Bleeding gums or periodontal disease

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of RiSE intervention: questionnaire | 8 weeks
  Feasibility of the RiSE intervention will be assessed at the end of the 8 week program. A written questionnaire will be completed by participants and asking participants to rate their level of satisfaction with the program on a scale of 0 to 10 with 0 being not satisfied at all to 10 being most satisfied. In addition, we will track class attendance and attrition rate.
Coping | 8 weeks
  Participants will complete written questionnaires at baseline, 4 weeks, and 8 weeks:
  Adaptive Coping. The Ways of Coping Checklist- Revised (WCCL-R) will be used to measure adaptive and non-adaptive coping. This is a 4-point Likert scale (0 to 3 ) that required the respondent to focus on a current stressor and to choose frequency of each of 66 proposed coping strategies. The WCCL-R is comprised of 5 subscales (scores are summed for each subscale) with higher scores indicating higher levels of the attribute measured by the subscale:
  Confrontational coping (scores range from 0 to 18) Distancing (scores range from 0 to 18) Self-controlling (scores range from 0 to 21) Seeking social support (scores range from 0 to 18) Accepting responsibility (scores range from 0 to 12) Escape-avoidance (scores range from 0 to 24) Planful problem-solving (scores range from 0 to 15) Positive reappraisal (scores range from 0 to 21)
Coping with Discrimination | 8 weeks
  Coping with Discrimination. The Coping with Discrimination Scale (CDS) is a 25-item scale that assesses coping strategies with discrimination. Items are answered using a 6-point Likert scale format ranging from strongly agree to strongly disagree. Scores are calculated for 5 subscales: Education/advocacy, Internalization, Drug/alcohol use, Resistance, and Detachment. Mean scores for each subscale range from 1 to 6 with higher scores indicating higher presence of the attribute measured.
Resilience | 8 weeks
  Resilience. The Connor-Davidson Resilience Scale- 25 will be used to measure resilience. The Connor Davidson Resilience Scale-25 is a 25 item questionnaire that examines the extent to which statements representing resilience, such as " I am able to adapt when changes occur" are true for the subject. Each item is evaluated on a five point Likert scale ranging from 0-4: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). Scores for items are summed and result in total score between 0-100 with higher scores indicating higher resilience.

SECONDARY OUTCOMES:
Inflammatory burden | 8 weeks
  Inflammatory burden will be measured at baseline and 8 weeks.
  Cytokine. ELISA will be used to measure circulating interleukin-6 (IL-6) (R & D Systems, Minneapolis MN). Sensitivity is < 0.7 pg/ml for IL-6. Intra assay variability is <7 %. Circulating IL-6 will be collected at baseline and 8 wks in both the intervention and control groups. Labs will be centrifuged for 7 minutes and frozen at -80 C for later batch analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Saban, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Wong MD, Shapiro MF, Boscardin WJ, Ettner SL. Contribution of major diseases to disparities in mortality. N Engl J Med. 2002 Nov 14;347(20):1585-92. doi: 10.1056/NEJMsa012979. PMID 12432046
- [Background] Wagner J, Abbott G. Depression and depression care in diabetes: relationship to perceived discrimination in African Americans. Diabetes Care. 2007 Feb;30(2):364-6. doi: 10.2337/dc06-1756. No abstract available. PMID 17259510
- [Background] Belgrave FZ, Abrams JA. Reducing disparities and achieving equity in African American women's health. Am Psychol. 2016 Nov;71(8):723-733. doi: 10.1037/amp0000081. PMID 27977253
- [Background] Mouton CP, Hayden M, Southerland JH. Cardiovascular Health Disparities in Underserved Populations. Prim Care. 2017 Mar;44(1):e37-e71. doi: 10.1016/j.pop.2016.09.019. PMID 28164826
- [Background] Wagner J, Lampert R, Tennen H, Feinn R. Exposure to Discrimination and Heart Rate Variability Reactivity to Acute Stress among Women with Diabetes. Stress Health. 2015 Aug;31(3):255-62. doi: 10.1002/smi.2542. Epub 2013 Nov 6. PMID 24194397
- [Background] Mwendwa DT, Sims RC, Madhere S, Thomas J, Keen LD 3rd, Callender CO, Campbell AL Jr. The influence of coping with perceived racism and stress on lipid levels in African Americans. J Natl Med Assoc. 2011 Jul;103(7):594-601. doi: 10.1016/s0027-9684(15)30385-0. PMID 21999034
- [Background] Wyatt SB, Williams DR, Calvin R, Henderson FC, Walker ER, Winters K. Racism and cardiovascular disease in African Americans. Am J Med Sci. 2003 Jun;325(6):315-31. doi: 10.1097/00000441-200306000-00003. PMID 12811228
- [Background] Williams DR, Jackson PB. Social sources of racial disparities in health. Health Aff (Millwood). 2005 Mar-Apr;24(2):325-34. doi: 10.1377/hlthaff.24.2.325. PMID 15757915
- [Background] Paradies Y. A systematic review of empirical research on self-reported racism and health. Int J Epidemiol. 2006 Aug;35(4):888-901. doi: 10.1093/ije/dyl056. Epub 2006 Apr 3. PMID 16585055
- [Background] Sutin AR, Stephan Y, Carretta H, Terracciano A. Perceived discrimination and physical, cognitive, and emotional health in older adulthood. Am J Geriatr Psychiatry. 2015 Feb;23(2):171-9. doi: 10.1016/j.jagp.2014.03.007. Epub 2014 Mar 21. PMID 24745563
- [Background] Todorova IL, Falcon LM, Lincoln AK, Price LL. Perceived discrimination, psychological distress and health. Sociol Health Illn. 2010 Sep;32(6):843-61. doi: 10.1111/j.1467-9566.2010.01257.x. Epub 2010 Jul 23. PMID 20649891
- [Background] Utsey SO, Payne YA, Jackson ES, Jones AM. Race-related stress, quality of life indicators, and life satisfaction among elderly African Americans. Cultur Divers Ethnic Minor Psychol. 2002 Aug;8(3):224-33. doi: 10.1037/1099-9809.8.3.224. PMID 12143100